CLINICAL TRIAL: NCT00418665
Title: A Randomized, Double Blind, Placebo Controlled Study Evaluating the Efficacy and Safety of AMG 531 Treatment of Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS) Receiving Lenalidomide.
Brief Title: A Safety and Efficacy Study to Evaluate AMG 531 Treatment in Subject With Myelodysplastic Syndrome Receiving Revlimid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20060102
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Myelodysplastic Syndromes; Thrombocytopenia
Keywords: Revlimid; Lenalidomide; Low Platelet Count; Low Risk Myelodysplastic Syndrome; Intermediate 1 Myelodysplastic Syndrome; MDS; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 750 mcg AMG 531 (Active Comparator): 750 μg AMG 531 weekly by subcutaneous injection + lenalidomide (10 mg orally per day) for 16 weeks (Part A)
  Interventions: Biological: AMG 531
- Placebo Part B (Placebo Comparator): Placebo weekly via subcutaneous injection + lenalidomide (10 mg orally per day) for 16 weeks (Part B)
  Interventions: Drug: Placebo
- Placebo Part A (Placebo Comparator): Placebo weekly via subcutaneous injection + lenalidomide (10 mg orally per day) for 16 weeks (Part A)
  Interventions: Drug: Placebo
- 500 mcg AMG 531 (Active Comparator): 500 μg AMG 531 weekly by subcutaneous injection + lenalidomide (10 mg orally per day) for 16 weeks (Part A)
  Interventions: Biological: AMG 531
- 750 mcg AMG531 Part B (Active Comparator): 750 μg AMG 531 biweekly by subcutaneous injection + lenalidomide (10 mg orally per day) for 16 weeks (Part B)
  Interventions: Biological: AMG 531

INTERVENTIONS:
Biological: AMG 531 — AMG 531 will be administered by subcutaneous injection at a dose of 500 or 750 μg.
  Arms: 500 mcg AMG 531; 750 mcg AMG 531; 750 mcg AMG531 Part B
Drug: Placebo — Subjects in the control group will receive placebo via subcutaneous injection.
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
This is a dose and schedule finding study of AMG 531 designed to assess the activity of AMG 531 to reduce the rate of clinically significant bleeding and blood transfusions in subjects with myelodysplastic syndrome (MDS) receiving lenalidomide. Subjects with MDS that are planned to receive at least four cycles of lenalidomide for treatment of their disease are appropriate to screen for this study.

All subjects meeting the eligibility criteria will receive lenalidomide 10 mg capsule by mouth daily every day of each 28-day cycle. Subjects will receive AMG 531 or placebo once a week by subcutaneous injection for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS by bone marrow biopsy based on the World Health Organization (WHO) classification
* Low or Intermediate-1 risk category MDS using the IPSS
* Planned to receive lenalidomide 10 mg capsule by mouth daily for all 28 days of each cycle for at least 4 cycles
* Eastern Cooperative Oncology (ECOG) performance status of 0-2
* Subjects must be at least 18 years of age or older

Exclusion Criteria:

* Prior exposure to >3 cycles of lenalidomide
* Exposure to lenalidomide within the last 30 days
* Prior history of leukemia or aplastic anemia
* Prior history of stem cell transplantation
* Prior malignancy (other than in situ cervical cancer or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for 3 years before randomization
* Active or uncontrolled infections
* Unstable angina, congestive heart failure [NYHA > class II], uncontrolled hypertension [diastolic > 100 mmHg], uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction
* History of arterial thrombosis ( eg, stroke or transient ischemic attack) in the past year
* History of venous thrombosis in the past year
* Received IL-11 within 4 weeks of screening
* Less than 4 weeks since receipt of any investigational drug or device
* Have previously received any other thrombopoietic growth factor
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* Known hypersensitivity to any recombinant E coli-derived product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Wang ES, Lyons RM, Larson RA, Gandhi S, Liu D, Matei C, Scott B, Hu K, Yang AS. A randomized, double-blind, placebo-controlled phase 2 study evaluating the efficacy and safety of romiplostim treatment of patients with low or intermediate-1 risk myelodysplastic syndrome receiving lenalidomide. J Hematol Oncol. 2012 Nov 29;5:71. doi: 10.1186/1756-8722-5-71. PMID 23190430
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 March 2007 through 24 July 2008
Groups:
- Placebo: Placebo weekly via subcutaneous injection plus lenalidomide 10 mg orally once per day for 16 weeks
- Romiplostim (AMG 531) 500 μg: Romiplostim (AMG 531) 500 μg weekly by subcutaneous injection plus lenalidomide 10 mg orally once per day for 16 weeks
- Romiplostim (AMG 531) 750 μg: Romiplostim (AMG 531) 750 μg weekly by subcutaneous injection plus lenalidomide 10 mg orally once per day for 16 weeks
Period: Treatment Period
Arm/Group | Placebo | Romiplostim (AMG 531) 500 μg | Romiplostim (AMG 531) 750 μg
Started | 12 | 14 | 13
Received Study Medication | 11 | 13 | 13
Completed | 7 | 8 | 9
Not Completed | 5 | 6 | 4
Not completed — Ineligibility determined | 1 | 1 | 0
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Requirement for alternative therapy | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 3
Period: Treatment Extension
Arm/Group | Placebo | Romiplostim (AMG 531) 500 μg | Romiplostim (AMG 531) 750 μg
Started | 7 | 8 | 9
Completed | 1 | 4 | 7
Not Completed | 6 | 4 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Requirement for alternative therapy | 2 | 2 | 0
Not completed — Physician Decision | 2 | 2 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Romiplostim 500 μg: Romiplostim (AMG 531) 500 μg weekly by subcutaneous injection plus lenalidomide 10 mg orally once per day for 16 weeks
- Romiplostim 750 μg: Romiplostim (AMG 531) 750 μg weekly by subcutaneous injection plus lenalidomide 10 mg orally once per day for 16 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Romiplostim 500 μg | Romiplostim 750 μg | Total
Number analyzed (Participants) | 12 | 14 | 13 | 39
Age Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (15.0) | 72.9 (11.4) | 66.7 (9.4) | 70.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 15
  Male | 8 | 8 | 8 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 11 | 13 | 12 | 36
  Black or African American | 0 | 0 | 1 | 1
  Hispanic or Latino | 1 | 1 | 0 | 2
International Prognostic Scoring System (IPSS) Score [Number; unit: Participants] — IPSS scoring for risk of myelodysplastic syndrome: 0 = low, 0.5 - 1.0 = intermediate 1, 1.5 - 2.0 = intermediate 2, ≥ 2.5 = high
  Participants
    0 | 4 | 4 | 6 | 14
    0.5 | 3 | 6 | 4 | 13
    1.0 | 3 | 2 | 3 | 8
    >1.0 | 1 | 1 | 0 | 2
    Missing | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a Clinically Significant Thrombocytopenic Event
Description: Occurrence of one or more clinically significant thrombocytopenic events, defined as either Common Terminology Criteria for Adverse Events (CTCAE) v. 3 grade 3 or 4 thrombocytopenia starting from week 3 of cycle 1 or receipt of platelet transfusions starting from week 1 of cycle 1 and continuing through the end of treatment visit.
Time Frame: Treatment period through interim follow-up visit (up to 16 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 500 μg | Romiplostim 750 μg
Number analyzed (Participants) | 12 | 14 | 13
Participants | 8 | 4 | 8
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 μg; Test type: Superiority or Other; Odds Ratio (OR) = 0.600, 95% CI [0.070 to 5.136] — Romiplostim/placebo
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 μg; Test type: Superiority or Other; Odds Ratio (OR) = 0.154, 95% CI [0.022 to 1.071] — Romiplostim/placebo

2. Secondary Outcome: Lenalidomide Dose Reduction and Delay Due to Thrombocytopenia
Description: Occurrence of lenalidomide dose reduction and delay due to thrombocytopenia
Time Frame: Treatment period (up to 16 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 500 μg | Romiplostim 750 μg
Number analyzed (Participants) | 12 | 14 | 13
Participants | 6 | 5 | 2
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 μg; Test type: Superiority or Other; Odds Ratio, log = 0.154, 95% CI [0.022 to 1.071] — Romiplostim/placebo
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 μg; Test type: Superiority or Other; Odds Ratio (OR) = 0.514, 95% CI [0.102 to 2.589] — Romiplostim/placebo

3. Secondary Outcome: Achieving an Overall Response (Complete Response (CR) or Partial Response (PR)) Determined by the Investigator Based on Modified International Working Group 2006 Response Criteria Guidelines
Description: CR = decrease in bone marrow blast (≤5%) and improvement in peripheral blood counts (Hgb ≥ 11 g/dL, platelets ≥ 100x10^9/L, neutrophils ≥ 1x10^9/L, peripheral blasts=0%). PR = improvement in peripheral blood counts plus a decrease in bone marrow blasts ≥50% but not ≤5, or decrease in International Prognostic Scoring System score.
Time Frame: Treatment period and post-treatment follow-up (up to 21 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 500 μg | Romiplostim 750 μg
Number analyzed (Participants) | 12 | 14 | 13
Participants | 1 | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 μg; Test type: Superiority or Other; Odds Ratio (OR) = 3.000, 95% CI [0.227 to 39.608] — Romiplostim/placebo
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 μg; Test type: Superiority or Other; Odds Ratio (OR) = 1.714, 95% CI [0.144 to 20.473] — Romiplostim/placebo

4. Secondary Outcome: Platelet Transfusion
Description: Occurrence of one or more platelet transfusions during the treatment period
Time Frame: Treatment period (up to 16 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 500 μg | Romiplostim 750 μg
Number analyzed (Participants) | 12 | 14 | 13
Participants | 4 | 4 | 4
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 μg; Test type: Superiority or Other; Odds Ratio (OR) = 0.911, 95% CI [0.097 to 8.529] — Romiplostim/placebo
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 μg; Test type: Superiority or Other; Odds Ratio (OR) = 0.866, 95% CI [0.175 to 4.278] — Romiplostim/placebo

ADVERSE EVENTS:
Time Frame: Up to 21 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Two subjects who were randomized to Placebo arm received one dose of Romiplostim inadvertently and were summarized in Romiplostim 750 mcg and 500 mcg arm, respectively.
Arm/Group | Placebo | Romiplostim 500 µg | Romiplostim 750 µg
Serious Adverse Events (participants affected / at risk) | 6/9 | 5/14 | 4/14
Other Adverse Events (participants affected / at risk) | 8/9 | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Romiplostim 500 µg (N=14) | Romiplostim 750 µg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Romiplostim 500 µg (N=14) | Romiplostim 750 µg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 5
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 4 | 8
Feeling cold (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 3 | 5 | 3
Pyrexia (General disorders) | 2 | 1 | 2
Ulcer haemorrhage (General disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Culture urine positive (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 3
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 4 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 5 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.